CLINICAL TRIAL: NCT00129532
Title: Randomized Controlled Trial of SAVVY and HIV in Ghana
Brief Title: Trial of SAVVY and HIV in Ghana
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biosyn (Industry)
Collaborators: FHI 360 (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9779
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2005-08

CONDITIONS: HIV Infections
Keywords: HIV transmission
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: 1.0% C31G SAVVY vaginal gel

SUMMARY:
Heterosexual contact is now the primary route of transmission for HIV worldwide. This study is a phase 3 trial designed to determine the effectiveness and safety of the 1.0% C31G (SAVVY) vaginal gel for the prevention of male-to-female transmission of HIV among women at high risk.

DETAILED DESCRIPTION:
Heterosexual contact is now the primary route of transmission for HIV worldwide. This study is a phase 3 multi-center, fully-masked, randomized, placebo controlled trial designed to determine the effectiveness and safety of the 1.0% C31G (SAVVY) vaginal gel for the prevention of male-to-female transmission of HIV among women at high risk.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 year old women
* HIV negative
* More than one sexual partner in past 3 months
* Average of 3 coital acts per week
* Willing to use vaginal gel and condoms for 12 months

Exclusion Criteria:

* HIV positive
* Pregnant

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2142
Dates: Start 2004-01

PRIMARY OUTCOMES:
combined incidence of HIV-1 and HIV-2

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Peterson, PhD, Study Chair — FHI 360
Locations (2):
- Ghana (2):
  - Noguchi Memorial Institute for Medical Research/University of Ghana, Accra
  - Komfo Anokye Teaching Hospital/Kwame Nkrumah University of Science and Technology, Kumasi

REFERENCES:
- [Derived] Peterson L, Nanda K, Opoku BK, Ampofo WK, Owusu-Amoako M, Boakye AY, Rountree W, Troxler A, Dominik R, Roddy R, Dorflinger L. SAVVY (C31G) gel for prevention of HIV infection in women: a Phase 3, double-blind, randomized, placebo-controlled trial in Ghana. PLoS One. 2007 Dec 19;2(12):e1312. doi: 10.1371/journal.pone.0001312. PMID 18091987